CLINICAL TRIAL: NCT05436288
Title: A Pilot Study of the Safety and Effectiveness of the EyeGate Ocular Bandage Gel, a 0.75% Crosslinked Hyaluronic Acid Applied Topically for the Improvement of Persistent Corneal Epithelial Defects (PED)
Brief Title: A Study of the KIO-201 (Ocular Bandage Gel) for Improving Persistent Corneal Epithelial Defects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kiora Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OBG PED-001
Record Dates: First submitted 2022-06-23; First posted 2022-06-29 (Actual); Results first posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Persistent Corneal Epithelial Defect

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single arm active (Experimental): KIO-201, a Crosslinked Thiolated Carboxymethyl Hyaluronic Acid 0.75% (CMHA-S), up to 6 times a day for 4 weeks.
  Interventions: Drug: KIO-201, a Crosslinked Thiolated Carboxymethyl Hyaluronic Acid 0.75% (CMHA-S)

INTERVENTIONS:
Drug: KIO-201, a Crosslinked Thiolated Carboxymethyl Hyaluronic Acid 0.75% (CMHA-S) — KIO-201 is a stand-alone drug therapy that acts as a barrier that minimizes mechanical lid friction and mechanically protects the ocular surface thereby reducing repeat injury and providing an environment that enables the body to repair the ocular surface whether the corneal epithelial defects are large or small.

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of topical KIO-201 in patients with persistent corneal epithelial defects (PED). KIO-201 will be administered six (6) times per day while awake for 4 weeks.

The primary exploratory effectiveness outcome for this study is the percentage of patients achieving corneal healing as determined by corneal fluorescein staining and photos. The effectiveness endpoint will be evaluated by a reader using digital photography of fluorescein stained slit lamp photos and image analysis.

DETAILED DESCRIPTION:
This is a prospective, exploratory study in which up to 10 patients (up to 20 eyes [minimum of 10 eyes]) diagnosed with Stage 1 and Stage 2 PED (as defined by fluorescein staining of the cornea and refractory to one or more conventional non-surgical treatments of at least 2 weeks) will receive KIO-201 with a dosing regimen of six (6) times per day over 4 weeks.

Both eyes are to be included if both eyes meet inclusion criteria and both eyes will be treated with KIO-201.

Patients will followed for a 4 week study.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older.
* Patients with persistent corneal epithelial defects (PED) (Stage 1 and Stage 2 PED).
* Patients with PED in one or both eyes, at least one eye meeting all study criteria.
* Have PED of at least 2 weeks' duration refractory to one or more conventional non-surgical treatments for Stage 1 and Stage 2 PED (i.e., preservative-free artificial tears, gels or ointments; discontinuation of preserved topical drops).

Exclusion Criteria:

* Have any active ocular infection (bacterial, viral, fungal or protozoal) in the affected eye(s).
* Schirmer's test without anesthesia ≤ 3 mm/ 5 minutes in the affected eye(s).
* Patients who have received amniotic membrane transplantation and have not healed.
* Patients treated with a bandage contact lens but have not healed.
* Prior surgical procedure(s) for the treatment of PED in the affected eye(s).
* Patients with lid abnormalities.
* Corneal disease that may affect outcomes.
* Stage 3 PED.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2023-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Graue, M.D., Principal Investigator — Instituto de Oftalmología Fundación Conde de Valenciana
Locations (1):
- Instituto de Oftalmología Fundación Conde de Valenciana, Mexico City, Chimalpopoca 14 Colonia Obrera, Mexico

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Arm Active
Started | 10
Completed | 8
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm Active
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Mexico | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Achieving Corneal Healing (<0.5 mm2 Lesion Size) of the Persistent Corneal Epithelial Defect at 4 Weeks
Description: Determined by corneal fluorescein staining and the effectiveness endpoint will also be evaluated by a reader using digital photography of fluorescein stained slit lamp photos and image analysis.
Time Frame: 4 weeks
Population: Eight (8) eyes were evaluable Five (5) of 8 (62.5%) of the evaluable participants achieved the primary endpoint of healing (<0.5 mm2 lesion size) at the 4-week period
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Active
Number analyzed (Participants) | 8
Participants | 5

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Single Arm Active
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 4/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm Active (N=10)
Eye Discomfort (Eye disorders) | 2 (3)
Change in Vision (Eye disorders) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2022-08-02): https://cdn.clinicaltrials.gov/large-docs/88/NCT05436288/Prot_000.pdf